CLINICAL TRIAL: NCT03812939
Title: An Observational Study Investigating Recurrence Rates of Type I Gastric Neuroendocrine Tumors Treated With Long-acting Somatostatin Analogs
Brief Title: Recurrence Rates of Type I Gastric Neuroendocrine Tumors Treated With Long-acting Somatostatin Analogs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Jing-Nan Li, Head of Gastroenterology, Peking Union Medical College Hospital
Other Study IDs: ZS-1788
Record Dates: First submitted 2019-01-13; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Gastric NET
MeSH Terms: interventions — Octreotide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Octreotide — Patients will receive 6-12 monthly injections every 28 (+/- 3) days.

SUMMARY:
This study evaluates the efficacy of Long-acting Somastostatin analogs as treatment for type I gastric neuroendocrine tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of gastric neuroendocrine tumor.
* Clinical diagnosis of Type I gastric NET: neuroendocrine tumor arising from atrophic body gastritis (ABG diagnosis should be based on hypergastrinemia and histological confirmation of gastric body atrophy on multiple biopsies performed in gastric antrum and body).
* Previous esophagogastroduodenoscopy: all visible NETs resected with R0 margin, confirmed no visible gastric NETs left, multiple biopsies taken to evaluate gastric atrophy and ECL status.
* No tumor metastases confirmed by endoscopic ultrasonography, CT scan or somatostatin receptor scintigraphy.
* SSA therapy is recommended by physician for disease management, and has not yet begun.
* Written informed consent obtained prior to treatment to be consistent with local regulatory requirements.

Exclusion Criteria:

* Pathological grading as G3 NET (Ki-67>20%).
* Patients with a known hypersensitivity to somatostatin analogs.
* Known gallbladder or bile duct disease, acute or chronic pancreatitis.
* Known medical condition related with prolonged QT interval.
* Pregnant or lactating women.
* Patients with serious complicated infections, or nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this therapy.
* Patients with any concurrent active malignancy other than non-melanoma skin cancers or carcinoma-in-situ of the cervix. Patients with previous malignancies but without evidence of disease for > 5 years will be allowed to enter the trial.
* Patients with a history of non-compliance to medical regimens.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type I gastric NET patients from tertiary medical center
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 1 year

SECONDARY OUTCOMES:
Change in clinical symptoms | 6 months to 1 year
  Measured by a questionnaire, including whether the patient presents with dyspepsia, abdominal pain, cramps, bloating, nausea, vomiting, lack of appetite, facial flushing.
Concentration of serum Gastrin | 6 months to 1 year
  Concentration of serum Gastrin after 12 hours of fasting
Enterochromaffin-like cell (ECL) status | 6 months to 1 year
  Normal Hyperplasia: ECL cell proliferation with a diameter <150 μm, distinguished in: normal pattern/simple hyperplasia, linear, micronodular and adenomatoid hyperplasia.
  Dysplasia: ECL cell proliferation >150 but <500 μm. Type I gastric carcinoid: ECL proliferation >500 μm.
Presence of side-effects of Octreotide | 6 months to 1 year
  Measured by a questionnaire for patients and clinician's report. Including: hypersensitivity, endocrine disorders (abnormal thyroid functions), metabolism and nutrition disorders (abnormal blood glucose), headache, bradycardia or tachycardia, dyspnea, gastrointestinal disorders (diarrhea, abdominal pain, nausea, constipation, flatulence), hepatobiliary disorders, skin disorders, injection site reaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Delle Fave G, O'Toole D, Sundin A, Taal B, Ferolla P, Ramage JK, Ferone D, Ito T, Weber W, Zheng-Pei Z, De Herder WW, Pascher A, Ruszniewski P; Vienna Consensus Conference participants. ENETS Consensus Guidelines Update for Gastroduodenal Neuroendocrine Neoplasms. Neuroendocrinology. 2016;103(2):119-24. doi: 10.1159/000443168. Epub 2016 Jan 19. No abstract available. PMID 26784901
- [Background] Merola E, Sbrozzi-Vanni A, Panzuto F, D'Ambra G, Di Giulio E, Pilozzi E, Capurso G, Lahner E, Bordi C, Annibale B, Delle Fave G. Type I gastric carcinoids: a prospective study on endoscopic management and recurrence rate. Neuroendocrinology. 2012;95(3):207-13. doi: 10.1159/000329043. Epub 2011 Jul 30. PMID 21811050
- [Background] Solcia E, Bordi C, Creutzfeldt W, Dayal Y, Dayan AD, Falkmer S, Grimelius L, Havu N. Histopathological classification of nonantral gastric endocrine growths in man. Digestion. 1988;41(4):185-200. doi: 10.1159/000199786. PMID 3072229